CLINICAL TRIAL: NCT06723171
Title: A 4-Week, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of the RXR Agonist Compound IRX4204 for the Treatment of Mild to Moderate Plaque Psoriasis
Brief Title: Evaluation of Safety and Efficacy of IRX4204 in Mild to Moderate Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Io Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRX4204Psoriasis201
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis; Plaque Type Psorisis; Plaque Psoriasis
Keywords: RXR; Psoriasis; plaque psoriasis; plaques; mild psoriasis; IRX4204; IO Therapeutics
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid | interventions — IRX4204; AGN 194204

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): IRX4204
  Interventions: Drug: IRX4204
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IRX4204 — Active Treatment
  Other Names: IRX4204Psoriasis; NRX194204
  Arms: Treatment
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if IRX4204 works to treat plaque psoriasis in adults. It will also learn about the safety of IRX4204. The main questions it aims to answer are:

* Does IRX4204 treat plaque psoriasis symptoms?
* Does IRX4204 treat plaque psoriasis symptoms better than someone who is not being treated?
* What medical problems do participants have when taking IRX4204?

Researchers will compare IRX4204 to a placebo (a look-alike substance that contains no drug) to see if the drug works to treat mild to moderate plaque psoriasis.

Participants will:

* Take IRX4204 every day for 28 days
* Visit the clinic once every week for checkups and tests
* Complete specific assessments about plaque psoriasis and changes to plaques

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Have a diagnosis of plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before the first administration of study treatment
3. Meet the following disease severity criteria for moderate to severe plaque psoriasis at Screening and Baseline visits:

   1. IGA Score of 3 or 4 AND
   2. Total affected body surface area of >3 to 10% for moderate and 10% to 15% for severe psoriasis
   3. Excludes participants with scalp only plaques
4. Be inadequately controlled with or intolerant of at least one prior topical therapy including but not limited to: corticosteroids, retinoids, vitamin D, vitamin D/steroid and retinoid/steroid combinations, tacrolimus, pimecrolimus, anthralin/dithranol, coal tar preparations, tapinarof, roflumilast for the treatment of psoriasis at both Screening and Baseline visits
5. In the opinion of the Investigator, be a candidate for phototherapy or systemic treatment for psoriasis
6. Completed appropriate washouts for prior treatments for psoriasis
7. Be considered, in the opinion of the Investigator, suitable candidates for RXR agonist therapy
8. Women participants of childbearing potential (WOCBP) (see Section 8.1.10) or sexually active male participants with partners of childbearing potential agree to practice a highly effective method of contraception (failure rate of < 1% per year when used consistently and correctly; see Section 8.1.10.1) prior to receiving, while receiving, and for at least 6 months after receiving the last administration of study intervention
9. WOCBP must have a negative highly sensitive serum beta-human chorionic gonadotropic (b-hCG) pregnancy test at Screening and confirmed at Baseline prior to receiving the first administration of study drug
10. WOCBP must agree not to donate eggs (ova, oocytes) or freeze for future and males must agree not to donate sperm for the purpose of reproduction for at least 6 months after receiving the last administration of study intervention.
11. Female participants must agree to not breastfeed while enrolled in this study and within 6 months after the last dose of study intervention
12. Sign an informed consent form (ICF) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study
13. Be willing to and able to adhere to the requirements in this protocol

Exclusion Criteria:

1. Has more than 15% of total body surface area affected by psoriasis plaques
2. Has a non-plaque form of psoriasis (e.g., erythrodermic, guttate, or pustular) at Screening or at time of randomization
3. Has current drug-induced psoriasis (e.g., a new onset of psoriasis or an exacerbation of psoriasis from beta-blockers, calcium channel blockers, or lithium)
4. Has confounding diagnoses including but not limited to palmoplantar pustulosis, eczematous dermatitis, contact/irritant dermatitis, acquired keratoderma
5. Has received within 12 weeks of the first dose (Day 1) any prior biologic (or biosimilars of) for the treatment of psoriasis, psoriatic arthritis, or any other indications that could impact the assessment of psoriasis. Prior biologic therapy includes but is not limited to TNF-inhibitors, IL-17 inhibitors, IL-12/23 inhibitors, IL-23 inhibitors
6. Has received within 4 weeks of the first dose (Day 1) any systemic immunosuppressives for the treatment of psoriasis or psoriatic arthritis, or any other indications that could impact the assessment of psoriasis, Phototherapy or narrow band laser (e.g., Excimer or XTRAC), lithium, antimalarials, or intramuscular (IM) gold. Systemic immunosuppressive therapy includes but is not limited to methotrexate, azathioprine, cyclosporine, JAK/TYK pathway inhibitors, 6-thioguanine, mercaptopurine, mycophenolate mofetil, tacrolimus, acitretin, or anakinra
7. Has received within 2 weeks of the first dose (Day 1) any topical medications for psoriasis or other conditions that could impact assessment of psoriasis, including but not limited to topical corticosteroids, retinoids, vitamin D analogs, combinations of calcipotriene and topical corticosteroids, tacrolimus, pimecrolimus, anthralin/dithranol, coal tar preparations, PDE4 inhibitors (e.g. crisaborole), or other topicals used for the treatment of psoriasis (tapinarof, roflumilast etc.)
8. Has received within 12 weeks or 5 half-lives (whichever is longer) of the first dose (Day 1) other biologic therapy or experimental antibody, any agent that modulates T-cells (e.g., natalizumab, abatacept etc.)
9. Has received within 4 weeks or 5 half-lives (whichever is longer) of the first dose (Day 1) any other experimental systemic therapy for any indication
10. Is currently enrolled in another study using an investigational agent or procedure
11. Has evidence of skin conditions that could interfere with clinical assessments of psoriasis (e.g. eczema, seborrheic dermatitis, or pityriasis rosea)
12. Has a current history of severe, uncontrolled or progressive systemic medical conditions including renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
13. Has unstable cardiovascular disease, defined as a recent clinical deterioration in the last 3 months (e.g., unstable angina, atrial fibrillation) or a cardiac hospitalization within the last 3 months
14. Currently has a known malignancy or has a history of malignancy within 5 years before screening with the exception of non-melanoma skin cancer curatively treated with no evidence of recurrence for at least 3 months before the first study drug administration or cervical carcinoma in situ of the cervix that has been treated with no evidence of recurrence for at least 3 years before the first study drug administration
15. Has a history of lymphoproliferative disease, including lymphoma, leukemia, monoclonal gammopathy, or signs/symptoms suggestive of possible lymphoproliferative disease
16. Has a transplanted organ (with the exception of a corneal transplant > 3 months before the first study drug administration)
17. Has unstable suicidal ideation or suicidal behavior, or a suicide attempt (including interrupted, aborted attempts and preparatory behaviors for suicide attempt), in the last 6 months
18. Has had a major surgery within 8 weeks of Screening or has such surgery planned during the time participant is expected to participate in the study
19. Has had a substance abuse problem within the previous 12 months
20. Has a history of chronic or recurrent infectious disease including but not limited to chronic renal infection, recurrent urinary tract infection (UTI), chronic respiratory infections (e.g., tuberculosis), skin infections, or fungal infections
21. Is currently being treated for a thyroid condition or have abnormalities in TSH, free T4 or T3 at Screening
22. Has had a serious infection (e.g., sepsis, pneumonia, pyelonephritis) requiring hospitalization within the 2 months before Screening
23. Has had herpes zoster (shingles) within 2 months prior to Screening
24. Has an active tuberculosis (TB) infection as confirmed by TB test during screening
25. Tests positive for hepatitis B virus (HBV) infection
26. Is seropositive for antibodies to hepatitis C virus (HCV). If the antibody test result is positive at screening, the participant will be allowed to be re-screened one time and enrolled after a negative HCV RNA test result
27. Is infected with human immunodeficiency virus (HIV)
28. Unable to avoid prolonged sun exposure or use of tanning beds or other ultraviolet light sources
29. Has received within 2 weeks of the first dose (Day 1) any prescribed anticoagulant, including but not limited to coumarins (such as warfarin), factor Xa inhibitors (i.e., apixaban, rivaroxaban), heparins (e.g., heparin, enoxaparin), and direct thrombin inhibitors
30. Has any condition that, in the opinion of the Investigator, would make participation not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments
31. Is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator
32. Any abnormal laboratory value greater than 2.5 times upper limit of normal (ULN). If one or more of the laboratory parameters is out of range, a single retest of laboratory values is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate if participants receiving IRX4204 achieve greater reduction in IGA scores when compared to participants receiving placebo | Baseline (Day 1) to Day 42
  Percentage of participants achieving an Investigator's Global Assessment (IGA) score of clear (0) or almost clear (1) at Day 28 with at least a 2-grade improvement from Baseline to end of study.

SECONDARY OUTCOMES:
To evaluate if participants receiving IRX4204 have greater improvement in participant reported outcomes when compared to participants receiving placebo | from Baseline (Day 1) to Day 28
  Change in Daily Quality of Life Index (DLQI) score will be evaluated. The DLQI is calculated by adding the score of each question, resulting in a minimum of 0 to a maximum of 30. The higher the score, the more quality of life is impaired.
To evaluate if participants receiving IRX4204 experience a greater reduction in affected Body Surface Area when compared to participants receiving placebo | from Baseline (Day 1) to Day 28
  Percent change in affected Body Surface Area (BSA) from Baseline to end of treatment will be evaluated. The body surface area refers to the total amount of skin on the body that is covered by psoriasis lesions and used to assess the severity of the condition. A higher percentage indicates a more severe case of psoriasis.
To evaluate if a greater proportion of participants receiving IRX4204 achieve PASI50, PASI75 and PASI90 when compared to participants receiving placebo | from Baseline (Day 1) to End of Study (Day 42)
  Proportion of participants to achieve PASI50 (50% or greater improvement from Baseline), PASI75, and PASI90 to the end of the study will be evaluated. Achieving PASI 50, PASI 75, and PASI 90 indicates different levels of improvement in psoriasis severity as measured by the Psoriasis Area and Severity Index (PASI) score, with PASI 50 indicating a 50% reduction from baseline, PASI 75 signifying a 75% reduction, and PASI 90 representing a 90% reduction in psoriasis symptoms. Higher PASI numbers signifying increasingly clearer skin.
To evaluate if participants receiving IRX4204 achieve greater improvement from baseline in disease and symptom severity as measured by the Psoriasis Area and Severity Index (PASI). | from Baseline (Day 1) to End of Treatment (Day 28)
  Change From Baseline to Day 28 in mean Psoriasis Area and Severity Index (PASI) score of participants receiving IRX4204 compared to placebo.

OTHER OUTCOMES:
Incidence of Treatment Emergent and Serious Adverse Events | from Baseline (Day 1) to End of Study (Day 42)
  The number of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs), and the number of participants who experienced TEAEs and SAEs will also be tabulated to evaluate the safety profile of IRX4204.

CONTACTS AND LOCATIONS:
Locations (1):
- Not posted, Webster, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided